CLINICAL TRIAL: NCT05973513
Title: Open Trial of Biofeedback for Respiratory Symptoms
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Natacha D. Emerson, Assistant Clinical Professor, University of California, Los Angeles
Other Study IDs: 21-000741-B
Record Dates: First submitted 2023-07-17; First posted 2023-08-03 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Shortness of Breath/Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Immediate Enrollment: We propose to study whether patients who complete a clinical six-session biofeedback protocol will demonstrate improvements in mental and physical health.

SUMMARY:
Biofeedback is a therapeutic paradigm that teaches patients how to gain awareness and control over previously unrecognized sympathetic changes such as body temperature, blood pressure, and heart rate. We propose to use a six session biofeedback protocol that includes heart-rate variability (HRV) biofeedback, respiration/relaxation training, and body temperature control to treat patients with unaddressed respiratory symptoms (e.g. shortness of breath) who are under the care of pulmonologists and have not responded to traditional biomedical approaches (e.g. inhalers, pulmonary rehab, etc.).

DETAILED DESCRIPTION:
Biofeedback is a therapeutic paradigm that teaches patients how to gain awareness and control over previously unrecognized sympathetic changes such as body temperature, blood pressure, and heart rate. Through a series of mind-body techniques, patients are taught to reduce sympathetic responses, leading to self-regulation over physiological responses that affect somatic sensitivity. The investigators propose to use a six session biofeedback protocol that includes heart-rate variability (HRV) biofeedback, respiration/relaxation training, and body temperature control to treat patients with unaddressed respiratory symptoms (e.g. shortness of breath) who are under the care of pulmonologists and have not responded to traditional biomedical approaches (e.g. inhalers, pulmonary rehab, etc.). The aim of the study is to determine whether patients who complete a six-session biofeedback protocol report a decrease in somatic symptoms, and improvements in self-rated mental health (depression, anxiety, quality of life) after the program and at three-months follow-up. The investigators will also study whether these improvements are also related to reduced healthcare utilization.

The investigators plan to recruit up to 100 participants in the study. Participants who are screened as eligible for biofeedback for their physical ailments or psychological complaints will be asked complete a set of questionnaires before, after, and three months' post-treatment to evaluate the utility of the biofeedback treatment protocol. These questionnaires will be available online and will be completed from home. Participants who are eligible to participate but cannot complete questionnaires from home will be given the option of completing the questionnaires in the office before the first biofeedback session. Participants that cannot be immediately enrolled in the protocol due to scheduling reasons will be asked to complete the questionnaires at recruitment to serve as wait-list controls. They will complete the same consent as other participants. The investigators anticipate that questionnaires will take 30 minutes to complete, totaling about 90 minutes for participants immediately enrolled and 120 minutes for wait-list controls.

Each biofeedback session will take 1 hour each. Session 1 of biofeedback will present the rationale and evidence for the treatment, teach breathing techniques, and introduce the biofeedback sensors for respiration, heart rate and temperature using the Biotrace software. The session will focus on breathing rate practice. Session 2 will introduce heart rate variability (HRV), cover breathing rhythm, and focus on the completion Resonance Frequency Assessment, an exercise to identify a participant's ideal breath rate for sustaining HRV. Session 3 will continue HRV practice using a separate software with video games, Alive. Session 4 will repeat session 3 but with more challenging practice of HRV video games. Session 5 will continue HRV practice in the first software (Biotrace) then will introduce participants to temperature control. Session 6 will repeat Session 5 but with more challenging practice for temperature control. Total time for participation will be approximately seven hours across three to six months.

ELIGIBILITY:
Inclusion Criteria:

1. participants must be between 18-60
2. English speaking
3. must have least one respiratory sx and have received care from a pulmonologist for this sx

Exclusion Criteria:

severe psychopathology (e.g., psychosis, active suicidality, moderate to severe intellectual impairment).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: (1) participants must be between 18-60; (2) English speaking; (3) must have least one respiratory sx and have received care from a pulmonologist for this sx
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in score on the PHQ-9 | After six week protocol and 3 months after six week protcol
  Improvement in self-rated depressive sx on the PHQ-9
Change in score on the GAD-7 | After six week protocol and 3 months after six week protcol
  Improvement in self-rated anxiety sx on the GAD-7
Change in score on the SF-36 | After six week protocol and 3 months after six week protcol
  Improvement in self-rated QOL on the SF-36
Change in score on the PHQ-15 | After six week protocol and 3 months after six week protcol
  Improvement in self-rated physical symptoms on the PHQ-15
Change in score on the PSQI | After six week protocol and 3 months after six week protcol
  Improvement in self-rated sleep quality and duration on the PSQI
Change in score on the St George's Respiratory Questionnaire (SGRQ) | After six week protocol and 3 months after six week protcol
  Improvement in self-rated respiratory sx on the SGRQ

SECONDARY OUTCOMES:
Change in healthcare utilization | After six week protocol and 3 months after six week protcol
  Reduced healthcare utilization: Fewer medical visits and use of prescription and OTC meds in last month

CONTACTS AND LOCATIONS:
Locations (1):
- Natacha Emerson, Los Angeles, California, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-07-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT05973513/ICF_000.pdf